CLINICAL TRIAL: NCT01062802
Title: Randomised Controlled Trial of Effect of Pre-operative Statin Use on Matrix Metalloproteinases (MMP) & Tissue Inhibitors of Matrix Metalloproteinases (TIMP) in Abdominal Aortic Aneurysm (AAA).
Brief Title: Statin Use in Abdominal Aortic Aneurysm Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CB/EL/R0135
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2007-12

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Statin group (Active Comparator)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80mg, once a day for four weeks.
  Arms: Statin group
Other: Placebo — Placebo given once daily for 4 weeks.
  Arms: Placebo

SUMMARY:
Aneurysm formation is associated with a chronic inflammatory response, depletion of smooth muscle cell population and excessive matrix metalloproteinases (MMPs) production. 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (statins) are lipid lowering agents with pleiotropic effects including anti-inflammatory activity. Elective open AAA repair patients will be randomised to receive either statin (Atorvastatin 80 mg) or placebo (dummy tablet) for 4 weeks pre-operatively. Tissue samples will be obtained from patient's aneurysm to assess MMP's and their inhibitors TIMP's. It is hypothesized that patients receiving statin will have reduced MMP's.

DETAILED DESCRIPTION:
All patients listed for elective open AAA repair will be screened for suitability to participate within the study. In this double blind randomized control trial patients will be recruited through vascular surgical outpatient clinics. After inclusion, informed consent and evaluation of base line characteristics patients will be given a prescription for study medication. This prescription was exchanged by the patient for medication at the hospital pharmacy. Randomization will be carried out by pharmacy with computer generated sequence with a sub group size of 4. This will ascertain the order of prescribed drug/ placebo. Pharmacy then dispensed the drug/ placebo in this order. Drug used will be Atorvastatin 80 mg, white, elliptical, film coated tablets debossed '80' on one side and 'PD 158' on the other side. The placebo is similar in shape and colour. Drug/ placebo will be given for 4 weeks pre-operatively. Full thickness infrarenal aortic samples will obtained at time of operation and the exact sample site will be recorded. Samples will be washed with 0.9% saline to remove blood and clots, snap-frozen and stored at -80C for subsequent MMP 2, 8 and 9 and TIMP 1 and 2 analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an AAA >5.5cm diameter listed for open AAA repair at least 3 weeks from screening attendance.

Exclusion Criteria:

* Patients already on statin,
* inability to provide informed written consent,
* contraindication to statin (intrinsic liver disease,
* chronic alcohol abuse, impaired renal function, unstable hypothyroidism,
* unexplained muscle aches, hypersensitivity to atorvastatin or any of its components),
* previous unilateral or bilateral lower limb amputation and concomitant use of fibrates,
* erythromycin,
* immunosuppressive drugs,
* antifungal drugs or lipid lowering drugs.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was the level of MMP-9 in aortic wall samples of patients on statins and placebo. | Sample obtained at time of operation

SECONDARY OUTCOMES:
The secondary outcome measures were the levels of MMP-2, MMP-8, TIMP-1, TIMP-2 and the variation in areas of peak wall stress due to statins. | Sample obtained at time of operation

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Chetter, MBChB, FRCS, Principal Investigator — Hull Royal Infirmary, Hull, United Kingdom.
Locations (1):
- Hull & east Yorkshire Hospitals NHS Trust, Hull, United Kingdom